CLINICAL TRIAL: NCT00002568
Title: A PHASE III RANDOMIZED STUDY OF CISPLATIN (NSC #119875) AND TAXOL (PACLITAXEL) (NSC #125973) WITH INTERVAL SECONDARY CYTOREDUCTION VERSUS CISPLATIN AND PACLITAXEL IN PATIENTS WITH SUBOPTIMAL STAGE III & IV EPITHELIAL OVARIAN CARCINOMA
Brief Title: Combination Chemotherapy With or Without Surgery in Treating Patients With Stage III Ovarian Epithelial Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000063600; GOG-152
Record Dates: First submitted 1999-11-01; First posted 2004-05-05 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2010-05

CONDITIONS: Ovarian Cancer
Keywords: stage III ovarian epithelial cancer; ovarian undifferentiated adenocarcinoma; ovarian mixed epithelial carcinoma; ovarian serous cystadenocarcinoma; ovarian mucinous cystadenocarcinoma; ovarian endometrioid adenocarcinoma; ovarian clear cell cystadenocarcinoma; Brenner tumor
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial; Brenner Tumor | interventions — Cisplatin; Paclitaxel

INTERVENTIONS:
Drug: cisplatin
Drug: paclitaxel
Procedure: conventional surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug or combining chemotherapy with surgery may kill more tumor cells.

PURPOSE: Randomized phase III trial to compare the effectiveness of combination chemotherapy consisting of paclitaxel and cisplatin with or without surgery in treating patients with stage III ovarian epithelial cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether secondary cytoreductive surgery improves the progression-free interval and survival in patients with suboptimally resected stage III ovarian epithelial carcinoma treated with paclitaxel/cisplatin. II. Determine the morbidity of secondary cytoreductive surgery in these patients. III. Assess prospectively the quality of life (QOL) of these patients and determine whether secondary cytoreductive surgery affects QOL.

OUTLINE: Randomized study. Following treatment on Regimen A, patients with stable or objective response are randomized to Arms I and II. Regimen A: 2-Drug Combination Chemotherapy. Paclitaxel (Bristol-Myers), Taxol, NSC-125973; Cisplatin, CDDP, NSC-119875. Arm I: Surgery followed by 2-Drug Combination Chemotherapy. Laparotomy with resection of residual disease; followed by Taxol/CDDP. Arm II: 2-Drug Combination Chemotherapy. Taxol; CDDP.

PROJECTED ACCRUAL: Approximately 470 patients will be entered over 20 months to provide 400 evaluable patients.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed primary ovarian epithelial cancer Stage III disease, i.e.: Greater than 1 cm residual intraperitoneal disease following exploratory laparotomy with maximum debulking Laparoscopic resection alone insufficient The following histologies are eligible: Serous adenocarcinoma Transitional cell carcinoma Mucinous adenocarcinoma Undifferentiated carcinoma Clear cell adenocarcinoma Mixed epithelial carcinoma Adenocarcinoma Endometrioid tumor Adenocarcinoma NOS Malignant Brenner's tumor No unclassified ovarian cancer (i.e., unexplored tumors thought to be of ovarian origin or tumors not verified as arising from ovarian stroma) No borderline (grade 0) or "probably malignant" carcinoma Measurable disease preferred Patients eligible for this protocol are also eligible for protocol GOG-136

PATIENT CHARACTERISTICS: Age: Any age Performance status: GOG 0-2 Hematopoietic: WBC at least 3,000/mm3 Absolute granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no more than 1.5 times normal ALT, AST, and GGT no more than 3 times normal Alkaline phosphatase no more than 3 times normal LDH no more than 3 times normal Renal: Creatinine no more than 2.0 mg/dL Cardiovascular: No history of congestive heart failure No myocardial infarction within 6 months No unstable angina Other: No septicemia or severe infection No acute hepatitis No severe gastrointestinal bleeding No second malignancy within 5 years except nonmelanomatous skin cancer Not pregnant or nursing Effective contraception required of fertile patients

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior cytotoxic chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy Surgery: See Disease Characteristics No more than 6 weeks since staging surgery

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 470 (Estimated)
Dates: Start 1994-06; Primary Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter G. Rose, MD, Study Chair — The Cleveland Clinic
Locations (55):
- United States (55):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - Women's Cancer Center, Palo Alto, California
  - Stanford University Medical Center, Stanford, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Lombardi Cancer Center, Georgetown University, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University School of Medicine, St Louis, Missouri
  - Cooper Hospital/University Medical Center, Camden, New Jersey
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Cancer Center of Albany Medical Center, Albany, New York
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - CCOP - Columbia River Program, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - CCOP - Baptist Cancer Institute, Memphis, Tennessee
  - Brookview Research, Inc., Nashville, Tennessee
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Cancer Center, University of Virginia HSC, Charlottesville, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Tacoma General Hospital, Tacoma, Washington

REFERENCES:
- [Background] von Gruenigen VE, Huang HQ, Gil KM, Gibbons HE, Monk BJ, Rose PG, Armstrong DK, Cella D, Wenzel L. A comparison of quality-of-life domains and clinical factors in ovarian cancer patients: a Gynecologic Oncology Group study. J Pain Symptom Manage. 2010 May;39(5):839-46. doi: 10.1016/j.jpainsymman.2009.09.022. PMID 20471545
- [Background] Farley JH, Tian C, Rose GS, Brown CL, Birrer M, Maxwell GL. Race does not impact outcome for advanced ovarian cancer patients treated with cisplatin/paclitaxel: an analysis of Gynecologic Oncology Group trials. Cancer. 2009 Sep 15;115(18):4210-7. doi: 10.1002/cncr.24482. PMID 19536873
- [Background] Winter WE 3rd, Maxwell GL, Tian C, Sundborg MJ, Rose GS, Rose PG, Rubin SC, Muggia F, McGuire WP; Gynecologic Oncology Group. Tumor residual after surgical cytoreduction in prediction of clinical outcome in stage IV epithelial ovarian cancer: a Gynecologic Oncology Group Study. J Clin Oncol. 2008 Jan 1;26(1):83-9. doi: 10.1200/JCO.2007.13.1953. Epub 2007 Nov 19. PMID 18025437
- [Background] Winter WE 3rd, Maxwell GL, Tian C, Carlson JW, Ozols RF, Rose PG, Markman M, Armstrong DK, Muggia F, McGuire WP; Gynecologic Oncology Group Study. Prognostic factors for stage III epithelial ovarian cancer: a Gynecologic Oncology Group Study. J Clin Oncol. 2007 Aug 20;25(24):3621-7. doi: 10.1200/JCO.2006.10.2517. PMID 17704411
- [Background] van der Burg ME, Vergote I; Gynecological Cancer Group of the EORTC. The role of interval debulking surgery in ovarian cancer. Curr Oncol Rep. 2003 Nov;5(6):473-81. doi: 10.1007/s11912-003-0008-8. PMID 14521806
- [Result] Wenzel L, Huang HQ, Monk BJ, Rose PG, Cella D. Quality-of-life comparisons in a randomized trial of interval secondary cytoreduction in advanced ovarian carcinoma: a Gynecologic Oncology Group study. J Clin Oncol. 2005 Aug 20;23(24):5605-12. doi: 10.1200/JCO.2005.08.147. PMID 16110020
- [Derived] Rose PG, Java JJ, Salani R, Geller MA, Secord AA, Tewari KS, Bender DP, Mutch DG, Friedlander ML, Van Le L, Method MW, Hamilton CA, Lee RB, Wenham RM, Guntupalli SR, Markman M, Muggia FM, Armstrong DK, Bookman MA, Burger RA, Copeland LJ. Nomogram for Predicting Individual Survival After Recurrence of Advanced-Stage, High-Grade Ovarian Carcinoma. Obstet Gynecol. 2019 Feb;133(2):245-254. doi: 10.1097/AOG.0000000000003086. PMID 30633128